CLINICAL TRIAL: NCT01199523
Title: A Phase 1, Randomized, Double-Blind, Placebo and Active Controlled, Parallel Crossover Study to Evaluate the Effect of Repeat Oral Doses of Mirabegron on Cardiac Repolarization in Healthy Male and Female Adult Subjects
Brief Title: A Study to Evaluate the Effect of Oral Mirabegron on the Heart in Healthy Males and Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 178-CL-077
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Subjects
Keywords: YM178; Mirabegron; QT
MeSH Terms: interventions — mirabegron; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- mirabegron high dose (Experimental)
  Interventions: Drug: mirabegron
- mirabegron medium dose (Experimental)
  Interventions: Drug: mirabegron
- mirabegron low dose (Experimental)
  Interventions: Drug: mirabegron
- moxifloxacin (Active Comparator)
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: Placebo — oral
  Arms: Placebo
Drug: mirabegron — oral
  Other Names: YM178
  Arms: mirabegron high dose; mirabegron low dose; mirabegron medium dose
Drug: moxifloxacin — oral
  Other Names: Avelox
  Arms: moxifloxacin

SUMMARY:
The objective of this study is to evaluate the effect of repeat oral dosing of mirabegron on ECG (electrocardiogram) measurements.

DETAILED DESCRIPTION:
Each subject will be randomized and participate in two 10-day treatment periods during which once daily dosing of mirabegron and mirabegron/moxifloxacin placebo or moxifloxacin and moxifloxacin/mirabegron placebo will occur followed by a 1-day post-treatment period. Each treatment period will be separated by a washout period of at least 12 days from the last dose of study drug on Day 10 of Period 1 to Day -4 of Period 2.

ELIGIBILITY:
Inclusion Criteria:

* The subject must weigh at least 45 kg and have a body mass index (BMI) between 20.0 and 28.5 kg/m2, inclusive
* The female subject must be post-menopausal (defined as at least 2 years without menses) or surgically sterile (at least 1 month prior to screening). All women of child bearing potential will be required to use adequate contraception consisting of two forms of birth control (one of which must be a barrier method), must not be lactating, and must not be breastfeeding during the study period and for 30 days after final study drug administration. All women of childbearing potential must have a negative serum pregnancy test. Male subjects with female spouses/partners who are of childbearing potential must use contraception consisting of two forms of birth control (one of which must be a barrier method) during the study period and for 30 days after final study drug administration.
* The subject must have negative test results for drugs of abuse and alcohol screens
* The subject must have good venous access

Exclusion Criteria:

* The subject is known to have hypersensitivity to mirabegron, or other adrenoreceptor agonists, or any of the constituents of the formulation used, or moxifloxacin or any member of the quinolone class of antimicrobial agents
* The subject has a history of syncope, cardiac arrest, cardiac arrhythmia or torsade de pointes, structural heart disease, valvular abnormalities, or family history of long QT syndrome
* The subject has experienced acute febrile illness within past 7 days
* The subject has a history of tendonitis and/or liver function abnormality related to quinolone antibiotic treatment
* The subject has a hyperthyroid disorder
* The subject has a history or presence of psychiatric illness, or any medical condition or disorder that may compromise evaluation of drug effect, or is incapable of being compliant with the study procedures
* The subject has donated or lost ≥ 450 mL blood within 56 days prior to study drug administration or has donated plasma within 7 days prior to study drug administration
* The subject has received or is anticipated to receive a prescription drug within 14 days prior to Day -4 of Period 1 (within 30 days prior to Day -4 of Period 1 for any long acting treatments such as depot formulations). Subject has taken any over-the-counter (OTC) medications, including complementary and alternative medicines (except for hormonal contraceptives not including depot formulations, hormone replacement therapy and occasional use of acetaminophen of up to 2000 mg/day but not more than 4 days per week) within 14 days prior to Day -4 of Period 1
* The subject has consumed alcohol, xanthine derivative-containing food/beverages (tea, chocolate), grapefruit juice, grapefruit-containing products or Seville oranges (e.g., bitter marmalade) within 48 hours before admission into the unit on Day -4 of Period 1
* The subject has a recent history of alcohol or other substance abuse or any history of alcohol or substance dependence (with the exception of nicotine). The subject consumes more than 5 units of alcoholic beverages per week
* The subject has used tobacco-containing products or nicotine-containing products within 6 months
* The subject is currently participating in another clinical trial or is taking or has been taking an investigational drug 30 days or 10 half lives (whichever is longer), prior to first study drug administration
* The subject is known to have hepatitis or human immunodeficiency virus (HIV)-1 and/or HIV-2, or is positive for hepatitis A antibody IgM, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody
* The subject has any skin condition likely to interfere with electrocardiographic electrode placement or adhesion
* The subject has a breast implant or a history of thoracic surgery likely to cause abnormality of the electrical conduction through thoracic tissues
* The subject is unable to tolerate a controlled, quiet study conduct environment, including avoidance during specified times (e.g., during ECG monitoring days) of music, TV, movies, games and activities that may cause excitement, emotional tension or arousal
* The subject is unwilling to comply with study rules, including attempting to void at restricted times (e.g., prior to ECG extraction windows), remaining quiet, awake, undistracted, motionless and supine during specified times, and avoiding vigorous exercise as directed

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
QTcl evaluated through electrocardiogram analysis | Day 1 to Day 11 in Treatment Period 1 and 2
  QTcI is a QT interval corrected for heart rate using individual-specific correction formula

SECONDARY OUTCOMES:
Pharmacodynamic assessment through electrocardiogram analysis | Day 1 to Day 11 in Treatment Period 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (2):
- United States (2):
  - Glendale, California
  - Baltimore, Maryland

REFERENCES:
- [Background] Malik M, van Gelderen EM, Lee JH, Kowalski DL, Yen M, Goldwater R, Mujais SK, Schaddelee MP, de Koning P, Kaibara A, Moy SS, Keirns JJ. Proarrhythmic safety of repeat doses of mirabegron in healthy subjects: a randomized, double-blind, placebo-, and active-controlled thorough QT study. Clin Pharmacol Ther. 2012 Dec;92(6):696-706. doi: 10.1038/clpt.2012.181. Epub 2012 Nov 14. PMID 23149929